CLINICAL TRIAL: NCT04344769
Title: Characterization of the Nrf2 Response in Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Maria V. Irazabal Mira, Principal Investigator, Mayo Clinic
Other Study IDs: 17-008806; R21DK118391 (NIH)
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Oxidative Stress; Antioxidant Response; Nrf2; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a previous diagnosis of ADPKD: Patients that have been diagnosed with ADPKD and meet the study's inclusion criteria
- Healthy individuals as controls: Age and gender-matched healthy controls

SUMMARY:
The purpose of this study is to characterize oxidative stress and the Nrf2 antioxidant response in early stages of Autosomal Dominant Polycystic Kidney Disease (ADPKD), while identifying candidate biomarkers.

DETAILED DESCRIPTION:
Intracellular Reactive Oxygen Species (ROS) concentration is a major determinant of cellular fate and is finely regulated by the cell's antioxidant systems. While low levels of ROS are required for pro-survival signaling, cell proliferation, growth, and energy metabolism, the excess of ROS or oxidative stress leads to inflammation, cell death, and disease/injury progression. Indeed, oxidative stress is commonly observed in several renal diseases including ADPKD. On the other hand, a surplus of antioxidants will not only neutralize ROS, but may result in the antithesis of oxidative stress, which is known as reductive stress. The Nuclear factor (erythroid-derived 2)-like 2 (Nrf2) is a transcription factor that integrates cellular stress signals and responds by regulating the expression of several antioxidant proteins. Activation of the Nrf2-mediated antioxidant defense pathway enhances ROS detoxification, conferring a more reduced intracellular environment that can promote cell survival and proliferation, a distinctive feature in ADPKD that underlies cyst formation and enlargement. Therefore, a better characterization of ROS levels and antioxidant response in ADPKD patients would allow development of more specific and effective therapies, while providing additional related biomarkers.

The investigators broad objective is to characterize oxidative stress and the Nrf2 antioxidant response in early stages of ADPKD, while identifying candidate biomarkers.

Participants in this study will have a blood and a urine sample collected to determine biomarkers of oxidative status and antioxidant response to study redox balance at early stages of the disease. In addition, an abdominal MRI will be performed to determine patient's total kidney volume (TKV).

ELIGIBILITY:
Inclusion Criteria (ADPKD Subjects):

* ADPKD (based on Ravine et al. criteria)
* Class 1 B-E according to our imaging classification
* Male and female subjects 18 - 30 years of age, inclusive
* Estimated GFR> 60 mL/min/m2 (CKD-EPI equation)
* Ability to provide written, informed consent.

Exclusion Criteria (ADPKD Subjects):

* Class 2 according to our imaging classification
* Concomitant systemic disease in the kidney (e.g. lupus, hepatitis B or C, amyloidosis)
* Diabetes mellitus (fasting glucose > 126 mg/dL or treatment with insulin or oral hypoglycemics).
* Predicted urine protein excretion in urinalysis >1 g/24 hrs
* Abnormal urinalysis suggestive of concomitant glomerular disease.
* Subjects having contraindications to, or interference with MRI assessments. [For example: ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, large abdominal/back tattoos, etc].
* Female subjects that are pregnant

Inclusion Criteria (Healthy Subjects):

* Male and female subjects 18 - 30 years of age, inclusive
* Estimated GFR> 60 mL/min/m2 (CKD-EPI equation)
* Ability to provide written, informed consent.

Exclusion Criteria (Healthy Subjects):

* Previous personal or family history of kidney disease.
* Concomitant systemic disease in the kidney (e.g. lupus, hepatitis B or C, amyloidosis)
* Diabetes mellitus (fasting glucose > 126 mg/dL or treatment with insulin or oral hypoglycemics).
* Presence of proteinuria
* Abnormal urinalysis suggestive glomerular disease.
* Subjects having contraindications to, or interference with MRI assessments. [For example: ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, large abdominal/back tattoos, etc]
* Female subjects that are pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female patients with a previous diagnosis of ADPKD that meet the inclusion criteria. In addition, patients will be matched 1:1 to age and gender healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Oxidative Status | Baseline
  Determination of common biomarkers of oxidative damage including but not limited to: 8-oxodeoxyguanosine, F2-isoprostanes, from urine and plasma samples
Assessment of Antioxidant Response | Baseline
  Determination of antioxidants including but not limited to: Heme Oxygenase 1 (HO-1), Superoxide dismutase (SOD), catalase, glutathione reductase (GSR), glutathione peroxidase (GPx), and NAD(P)H dehydrogenase [quinone] 1 (NOQ1), glutathione, Nrf2 from urine and plasma samples
Total kidney volume (TKV) | Baseline
  Determined by MRI

SECONDARY OUTCOMES:
Assessment of Kidney Injury | Baseline
  Determination of kidney injury biomarkers including but not limited to: Kidney Injury Molecule 1 (KIM-1), Neutrophil gelatinase-associated lipocalin (NGAL), Monocyte chemotactic protein-1 (MCP-1), Transforming growth factor-β1 (TGF-β1),

CONTACTS AND LOCATIONS:
Overall Officials: Maria V. Irazabal, M.D., Ph.D, Principal Investigator — Mayo Translational PKD Center, Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials